CLINICAL TRIAL: NCT01363700
Title: Double-masked, Comparison Study of DE-114 Ophthalmic Solution in Patients With Allergic Conjunctivitis - Phase 3, Confirmatory Study -
Brief Title: Study of DE-114 Ophthalmic Solution in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 01141101
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; Ophthalmic Solutions

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DE-114 ophthalmic solution
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo ophthalmic solution
- 3 (Active Comparator)
  Interventions: Drug: Olopatadine Hydrochloride 0.1% Ophthalmic Solution

INTERVENTIONS:
Drug: DE-114 ophthalmic solution
  Other Names: Epinastine ophthalmic solution
  Arms: 1
Drug: Placebo ophthalmic solution
  Arms: 2
Drug: Olopatadine Hydrochloride 0.1% Ophthalmic Solution
  Arms: 3

SUMMARY:
The purpose of the study is to demonstrate safety and efficacy of DE-114 ophthalmic solution compared to its Placebo and Olopatadine hydrochloride 0.1% ophthalmic solution in patients with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent.
* Has a positive result from an allergen-specific IgE antibody test.
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Ages: 20 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Primary Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Japan

REFERENCES:
- [Derived] Fujishima H, Ohashi Y, Takamura E. Efficacy of epinastine hydrochloride ophthalmic solution in allergic conjunctivitis by conjunctival cedar pollen allergen challenge. Ann Allergy Asthma Immunol. 2014 Oct;113(4):476-81. doi: 10.1016/j.anai.2014.07.007. Epub 2014 Aug 20. PMID 25163405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Period1 comparison with placebo (Epinastine vs Placebo)
  * Period2 comparison with olopatadine (Epinastine vs Olopatadine)
Pre-assignment Details: All participants completed Period 1 were randomized 1:1 to 2 groups in Period 2.
Groups:
- Epinastine / Placebo Period1; Epinastine / Placebo Period2: Epinastine / Placebo : Epinastine ophthalmic solution in one eye and vehicle of DE-114 ophthalmic solution in the other eye, Both eye received 1 drop at designated visits.
- Epinastine / Epinastine Period1: Epinastine / Epinastine : Epinastine ophthalmic solution, 1 drop in each eye at designated visits.
- Placebo / Placebo Period1: Placebo / Placebo : vehicle of DE-114 ophthalmic solution, 1 drop in each eye at designated visits.
- Olopatadine / Placebo Period2: Olopatadine / Placebo : Olopatadine ophthalmic solution in one eye and vehicle of DE-114 ophthalmic solution in the other eye, Both eye received 1 drop at designated visits.
Period: Epinastine vs Placebo Period1
Arm/Group | Epinastine / Placebo Period1 | Epinastine / Epinastine Period1 | Placebo / Placebo Period1 | Olopatadine / Placebo Period2 | Epinastine / Placebo Period2
Started | 43 | 22 | 22 | 0 (No Allocation) | 0 (No Allocation)
Completed | 43 | 21 | 22 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Epinastine vs Olopatadine Period2
Arm/Group | Epinastine / Placebo Period1 | Epinastine / Epinastine Period1 | Placebo / Placebo Period1 | Olopatadine / Placebo Period2 | Epinastine / Placebo Period2
Started | 0 (No Allocation) | 0 (No Allocation) | 0 (No Allocation) | 43 | 43
Completed | 0 | 0 | 0 | 43 | 43
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Epinastine / Placebo Period1: Epinastine / Placebo : DE-114 ophthalmic solution in one eye and vehicle of DE-114 ophthalmic solution in the other eye, Both eye received 1 drop at designated visits.
- Epinastine / Epinastine Period1: Epinastine / Epinastine : DE-114 ophthalmic solution, 1 drop in each eye at designated visits.
- Total: Total of all reporting groups
Arm/Group | Epinastine / Placebo Period1 | Epinastine / Epinastine Period1 | Placebo / Placebo Period1 | Total
Number analyzed (Participants) | 43 | 22 | 22 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.0) | 39.0 (10.0) | 39.7 (11.7) | 39.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — * After "Epinastine vs Placebo", allocate subjects to Olopatadine / Placebo or Epinastine / Placebo for "Epinastine vs Olopatadine".
  * Demographic statistics in whole periods were not analyzed.
  Participants
    Female | 17 | 11 | 11 | 39
    Male | 26 | 11 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Itching Score Compared to Placebo Period1
Description: A conjunctivitis allergic challenge (CAC) was performed 4 hours after drop instillation. Mean ocular itching score was assessed by the subject at 3, 5, and 10 min post challenge and graded on a 5 points scale of 0-4 where 0=no itching and 4=incapacitating itch. Count unit was defined each eye.
  The endpoint used the average score of three time points (3, 5, and 10 minutes) after allergen challenge .
Time Frame: Visit 5 (3, 5, and 10 minutes post-CAC)
Measure: Mean (Standard Error); unit: score
Groups:
- Epinastine (DE-114) Ophthalmic Solution; Placebo Ophthalmic Solution: Count unit was defined each eye.
Arm/Group | Epinastine (DE-114) Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 87 | 87
score | 0.4 (0.1) | 1.7 (0.1)
Statistical Analysis 1: Comparison: Epinastine (DE-114) Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.52 to -1.11]

2. Primary Outcome: Mean Hyperemia Score Compared to Placebo Period1
Description: A conjunctivitis allergic challenge (CAC) was performed 4 hours after drop instillation. Mean palpebral and bulbar conjunctiva hyperemia was assessed by the investigator at 5, 10, and 20 min post challenge and graded on a 4 points scale of 0-3 (0=none and 3= extremely severe). Total hyperemia score is defined as the sum of the palpebral and bulbar conjunctiva scores. Count unit was defined each eye.
  The endpoint used the average score of three time points (5, 10, and 20 minutes) after allergen challenge .
Time Frame: Visit 5 (5, 10, and 20 minutes post-CAC)
Measure: Mean (Standard Error); unit: score
Arm/Group | Epinastine (DE-114) Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 87 | 87
score | 2.7 (0.1) | 4.1 (0.2)
Statistical Analysis 1: Comparison: Epinastine (DE-114) Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.71 to -0.92]

3. Secondary Outcome: Mean Ocular Itching Score Compared to Olopatadine Period2
Description: A conjunctivitis allergic challenge (CAC) was performed 4 hours after drop instillation. Mean ocular itching score was assessed by the subject at 3, 5, and 10 min post challenge on a 5 points scale of 0-4 where 0=no itching and 4=incapacitating itch.
  The endpoint used the average score of three time points (3, 5, and 10 minutes) after allergen challenge .
Time Frame: Visit 7 (3, 5, and 10 minutes post-CAC)
Measure: Mean (Standard Error); unit: score
Groups:
- Olopatadine Ophthalmic Solution; Placebo Ophthalmic Solution: Count unit was defined each eye.
Arm/Group | Epinastine (DE-114) Ophthalmic Solution | Olopatadine Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 43 | 43 | 86
score | 0.2 (0.1) | 0.2 (0.1) | 1.5 (0.1)
Statistical Analysis 1: Comparison: Epinastine (DE-114) Ophthalmic Solution vs Olopatadine Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Non-Inferiority or Equivalence — Non-inferiority in Mean Ocular itching score compared to Olopatadine was assessed on the non-inferiority margin (0.5) with the upper limit of the confidence interval of the difference between the Epinastine (DE-114) and Olopatadine treatment groups; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.21 to 0.08]

4. Secondary Outcome: Mean Hyperemia Score Compared to Olopatadine Period2
Description: A conjunctivitis allergic challenge (CAC) was performed 4 hours after drop instillation. Mean palpebral and bulbar conjunctiva hyperemia was assessed by the investigator at 5, 10, and 20 min post challenge and graded on a 4 points scale of 0-3 (0=none and 3= extremely severe). Total hyperemia score is defined as the sum of the palpebral and bulbar conjunctiva scores.
  The endpoint used the average score of three time points (5, 10, and 20 minutes) after allergen challenge .
Time Frame: Visit 7 (5, 10, and 20 minutes post-CAC)
Measure: Mean (Standard Error); unit: score
Arm/Group | Epinastine (DE-114) Ophthalmic Solution | Olopatadine Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 43 | 43 | 86
score | 2.4 (0.2) | 2.7 (0.2) | 3.7 (0.1)
Statistical Analysis 1: Comparison: Epinastine (DE-114) Ophthalmic Solution vs Olopatadine Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Non-Inferiority or Equivalence — Non-inferiority in Mean Ocular hyperemia score compared to Olopatadine was assessed on the non-inferiority margin (0.5) with the upper limit of the confidence interval of the difference between the Epinastine (DE-114) and Olopatadine treatment groups; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.81 to 0.22]

ADVERSE EVENTS:
Groups:
- Epinastine (DE-114) Ophthalmic Solution Period1; Placebo Ophthalmic Solution Period1; Epinastine (DE-114) Ophthalmic Solution Period2; Olopatadine Ophthalmic Solution Period2; Placebo Ophthalmic Solution Period2: Count unit was defined each eye.
Arm/Group | Epinastine (DE-114) Ophthalmic Solution Period1 | Placebo Ophthalmic Solution Period1 | Epinastine (DE-114) Ophthalmic Solution Period2 | Olopatadine Ophthalmic Solution Period2 | Placebo Ophthalmic Solution Period2
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/87 | 0/43 | 0/43 | 0/86
Other Adverse Events (participants affected / at risk) | 0/87 | 0/87 | 0/43 | 0/43 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No